CLINICAL TRIAL: NCT00127296
Title: Comparison of the Accuracy and Precision of NovoLog® Mix 70/30 FlexPen® to Vial and Syringe in Patients With Type 2 Diabetes Mellitus
Brief Title: Reliability of Dosing With NovoLog® Mix 70/30 FlexPen® Compared With Vial and Syringe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BIASP-1654
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Syringes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: FlexPen®
Device: vial and syringe

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to compare desired (target) with actual target amounts of insulin dispensed using NovoLog® Mix 70/30 FlexPen® and vial and syringe in subjects with type 2 diabetes mellitus. No insulin is administered in this trial - insulin is dispensed into an empty vial.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Insulin naive
* No previous experience administering injections

Exclusion Criteria:

* Any condition that, in the Investigator and/or Sponsor's opinion, could interfere with the results of this trial

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-07; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Combined measure of accuracy and precision between target and measured amounts of insulin dispensed (mean square percent difference)

SECONDARY OUTCOMES:
Patient preference
Accuracy (mean relative error)
Precision (coefficient of variation)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, San Antonio, Texas, United States

REFERENCES:
- [Result] Schwartz S, Khutoryansky N, Braceras R. Comparison of resource utilisation, preference and handling of a pre-filled pen and vial/syringe in patients with type 2 diabetes mellitus. Journal of Clinical Research 2007; 10: 1-10
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com